CLINICAL TRIAL: NCT06066320
Title: A Comparison of Acute Psychobiological Responses to the Mannheim Multicomponent Stress Test and the Trier Social Stress Test
Brief Title: A Comparison of Acute Psychobiological Responses to Laboratory Stress Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Daniel Kashi, Postdoctoral Research Officer, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ORION study 1B
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Between subjects design to compare psychobiological responses in participants randomised to either the MMST or the TSST. Stratified block randomisation will be used to evenly distribute participants to the MMS or the TSST based upon sex (male or female) and trait anxiety (low STAI-T score <40 or high STAI-T score ≥40).
Who Masked: Participant
Masking Description: Participants will be unaware of the true nature of experimental trials until a final debrief scheduled after acute stress exposure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMST (Experimental)
  Interventions: Behavioral: MMST
- TSST (Active Comparator)
  Interventions: Behavioral: TSST

INTERVENTIONS:
Behavioral: MMST — Participants randomised to the MMST group will complete the computer based paced auditory serial addition task (PASAT-C) in the presence of one observer and is informed that incorrect answers result in reduced monetary compensation. Simultaneously, the participant is exposed to emotionally evocative images and white noise via headphones
  Arms: MMST
Behavioral: TSST — Participants randomly assigned to the TSST condition will be exposed to a traditional TSST protocol. The TSST consists of a preparation phase (5 min), followed by a mock job interview and a mental arithmetic task (5 min each) in front of a panel consisting of two observers and a video recording device.
  Arms: TSST

SUMMARY:
The Mannheim Multicomponent Stress Test (MMST) is a validated laboratory stress test that combines cognitive, emotional, acoustic and motivational stress components. However the utility of the MMST as a viable alternative to the more commonly used Trier social stress test (TSST) to elicit HPA reactivity remains unclear as meaningful increases in saliva cortisol (> 2.5 nmol/l) have been shown to occur in <50% of participants yet the TSST typically elicits meaningful increases in saliva cortisol in >70% of participants; likely as a consequence of the greater social evaluative component in the TSST.

Using a randomised between groups design, this study aims to compare psychobiological responses to the MMST and TSST.

ELIGIBILITY:
Inclusion Criteria:

Participants who…

* have read and signed the study informed consent
* are healthy, recreationally active men and women aged 18-35 years
* are willing to provide saliva samples throughout through the duration of the study
* are using monophasic birth control (women only)

Exclusion Criteria:

Participants who…

* have a recent history or are a current smoker
* are currently taking prescription/Over-the-counter medication (excluding females taking oral combined contraception
* consume ≥ 91 units of alcohol per month
* have a clinically diagnosed history of cardiovascular and/or metabolic disease including diabetes and abnormal blood pressure
* are pregnant
* have a recent or ongoing viral or bacterial illness in past 4 weeks
* have a clinically diagnosed psychiatric disorder
* have a clinically diagnosed sleeping disorder
* have a clinically diagnosed gambling addiction
* BMI ≥ 30 kg/m2 - calculated in the online health screening questionnaire
* Endurance trained or engage in ≥3.5 hours of physical activity a week

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Change in saliva cortisol (pre-post stress) | Change from 5 minutes pre to peak post stress test (MMST or TSST)
  Changes in the concentration of saliva free cortisol assessed by ELISA.

SECONDARY OUTCOMES:
State anxiety inventory (STAI-S) response to acute psychological stress | Change from 5 minutes pre to after stress challenge (immediately after acute psychological stress and 60 minutes after the test) will be compared.
  assessed using the state scale of the state trait anxiety inventory (STAI-S), consisting of a 20-item scale for measuring the intensity of anxiety as an emotional state (S-Anxiety). The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80)
Heart rate | Continuously assessed from 30 minutes before to 60 minutes after the stress tests and control tests
  Continuous measurement of heart rate will be assessed using a telemetric chest strap.
Salivary alpha amylase (sAA) | Change from 5 minutes pre to immediately post stress test
  a biomarker for stress-induced activity of the sympathetic nervous system (SNS), assessed by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Neil P Walsh, PHD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Faculty of Science, Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No